CLINICAL TRIAL: NCT01336205
Title: An Open-Label 52-week Study to Assess the Long-Term Safety of NKTR-118 in Opioid-Induced Constipation (OIC) in Patients With Non-Cancer-Related Pain
Brief Title: Assessment of Long-term Safety in Patients With Non-cancer-related Pain and Opioid-induced Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3820C00008
Record Dates: First submitted 2011-04-14; First posted 2011-04-15 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Opioid-Induced Constipation (OIC)
Keywords: Non-Cancer-Related Pain; Opioid-Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral Treatment
  Interventions: Drug: NKTR-118
- 2 (Active Comparator): Oral treatment
  Interventions: Drug: Usual care

INTERVENTIONS:
Drug: NKTR-118 — 25 mg oral tablet once daily
  Arms: 1
Drug: Usual care — As prescribed by the investigator
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of NKTR-118 treatment of opioid-induced constipation (OIC) in patients with non-cancer-related pain.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study-specific procedures.
* NEW PATIENTS ONLY: Self-reported active symptoms of OIC at screening (<3 SBMs/week and experiencing >1 reported symptom of hard/lumpy stools, straining, or sensation of incomplete evacuation/anorectal obstruction in at least 25% of the BMs over the previous 4 weeks); and Documented confirmed OIC (<3 SBMs/week on average over the 2-week OIC confirmation period.
* PATIENTS ENROLLING FROM OTHER NKTR-118 STUDIES: Receiving a stable maintenance opioid regimen consisting of a total daily dose of 30 mg to 1000 mg or oral morphine, or equianalgesic amount(s) of 1 or more opioid therapies.
* FOR PATIENTS RANDOMIZED TO RECEIVE NKTR-118: Willingness to stop all laxatives and other bowel regimens including prune juice and herbal products throughout the 52-week treatment period, and to use only bisacodyl as rescue medication if BM has not occurred within at least 72 hours of the last recorded BM.

Exclusion Criteria:

* Patients receiving Opioid regimen for treatment of pain related to cancer.
* History of cancer within 5 years from first study visit with the exception of basal cell cancer and squamous cell skin cancer.
* Medical conditions and treatments associated with diarrhea, intermittent loose stools, or constipation.
* Other issues related to the gastrointestinal tract that could impose a risk to the patient.
* Pregnancy or lactation.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 844 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, Study Director — AstraZeneca
Locations (169):
- United States (169):
  - Research Site, Athens, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Pell City, Alabama
  - Research Site, Garden Grove, Arizona
  - Research Site, Goodyear, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Tuscon, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, North Little Rock, Arkansas
  - Research Site, Sherwood, Arkansas
  - Research Site, Arcadia, California
  - Research Site, Chino, California
  - Research Site, Encino, California
  - Research Site, Fremont, California
  - Research Site, Garden Grove, California
  - Research Site, Huntington Park, California
  - Research Site, La Mesa, California
  - Research Site, Laguna Hills, California
  - Research Site, Lakewood, California
  - Research Site, Long Beach, California
  - Research Site, Oceanside, California
  - Research Site, Orange, California
  - Research Site, Pasadena, California
  - Research Site, Riverside, California
  - Research Site, San Bernardino, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Santa Ana, California
  - Research Site, Walnut Creek, California
  - Research Site, Whittier, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Bradenton, Florida
  - Research Site, Brooksville, Florida
  - Research Site, Chiefland, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, DeBary, Florida
  - Research Site, Deerfield Beach, Florida
  - Research Site, Delray Beach, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Eustis, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jackson, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Largo, Florida
  - Research Site, Lauderhill, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, North Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orange City, Florida
  - Research Site, Orlando, Florida
  - Research Site, Oviedo, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pinellas Park, Florida
  - Research Site, Plantation, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Saint Doral, Florida
  - Research Site, South Miami, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, West Palm, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Alpharetta, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Suwanee, Georgia
  - Research Site, Tucker, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Bloomington, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Schaumburg, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Council Bluffs, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Lansing, Kansas
  - Research Site, Overland Park, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Hollywood, Maryland
  - Research Site, Pikesville, Maryland
  - Research Site, Reisterstown, Maryland
  - Research Site, Watertown, Massachusetts
  - Research Site, Calamazoo, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Fremont, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Clifton, New Jersey
  - Research Site, Freehold, New Jersey
  - Research Site, Lumberton, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Willingboro, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Great Neck, New York
  - Research Site, Hartsdale, New York
  - Research Site, New York, New York
  - Research Site, North Massapequa, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Elkin, North Carolina
  - Research Site, Flat Rock, North Carolina
  - Research Site, Harrisburg, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, Morrisville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Beavercreek, Ohio
  - Research Site, Centerville, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Downingtown, Pennsylvania
  - Research Site, Jenkintown, Pennsylvania
  - Research Site, Norristown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pottstown, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Clarksville, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Milan, Tennessee
  - Research Site, New Tazewell, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Hurst, Texas
  - Research Site, Lexington, Texas
  - Research Site, Marshall, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugarland, Texas
  - Research Site, Victoria, Texas
  - Research Site, Clinton, Utah
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, St. George, Utah
  - Research Site, West Jordan, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Springfield, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Middleton, Wisconsin

REFERENCES:
- [Derived] Webster L, Chey WD, Tack J, Lappalainen J, Diva U, Sostek M. Randomised clinical trial: the long-term safety and tolerability of naloxegol in patients with pain and opioid-induced constipation. Aliment Pharmacol Ther. 2014 Oct;40(7):771-9. doi: 10.1111/apt.12899. Epub 2014 Aug 12. PMID 25112584
- See also: Clinical_Study_Report_Synopsis_D3820C00008 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1390&filename=Clinical_Study_Report_Synopsis_D3820C00008.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in the United States between 18 April 2011 and 03 December 2012.
Pre-assignment Details: The study duration was 54 to 58 weeks. New patients underwent an initial screening period lasting up to 2 weeks and a 2-week OIC confirmation period. New patients and patients enrolling from another study (also referred to as 'roll over patients') entered the 52-week treatment period, followed by a 2 week follow-up period.
Groups:
- NKTR-118 25 mg: NKTR-118 25 mg QD, oral treatment
- Usual Care: Laxative treatment regimen for OIC determined by the investigator according to his/her best clinical judgment.
Period: Overall Study
Arm/Group | NKTR-118 25 mg | Usual Care
Started | 563 | 281
Completed | 330 | 192
Not Completed | 233 | 89
Not completed — Other | 22 | 9
Not completed — Lost to Follow-up | 40 | 20
Not completed — Study-Specific Withdrawal Criteria | 16 | 7
Not completed — Lack of Efficacy | 4 | 0
Not completed — Severe noncompliance with protocol | 9 | 2
Not completed — Adverse Event | 56 | 6
Not completed — Death | 1 | 1
Not completed — Eligibility Criteria Not Fulfilled | 9 | 6
Not completed — Withdrawal by Subject | 72 | 38
Not completed — Did not receive treatment | 4 | 0

BASELINE CHARACTERISTICS:
Population: A total of 36 patients (11 patients in the Usual Care group and 25 new patients in the NKTR-118 25 mg group) had either: a) previously or concurrently participated in the NKTR-118 program at another study center; or b) were randomized at sites where data integrity issues were identified. These patients were excluded from the Safety analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | NKTR-118 25 mg | Usual Care | Total
Number analyzed (Participants) | 534 | 270 | 804
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (10.09) | 52.7 (10.24) | 52.7 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 353 | 179 | 532
  Male | 181 | 91 | 272
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 423 | 204 | 627
  Black or African American | 98 | 60 | 158
  Asian | 4 | 3 | 7
  American Indian or Alaska Native | 4 | 1 | 5
  Other | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Patients Experiencing at Least One Adverse Event (AE)
Description: The incidence of patients experiencing at least one AE during the randomized treatment and follow-up periods was calculated.
Time Frame: Baseline (Week 0) to end of the follow-up period
Population: The Safety analysis set included all randomized patients who received at least 1 dose of IP and patients who received Usual Care, with the exception of patients who were randomized multiple times within the program at different centers or patients who were randomized at sites where data integrity issues were identified.
Measure: Number; unit: Participants
Arm/Group | NKTR-118 25 mg | Usual Care
Number analyzed (Participants) | 534 | 270
Participants | 437 | 195

2. Primary Outcome: Incidence of Patients Experiencing AEs That Resulted in Discontinuation of Investigational Product (IP)
Description: The incidence of patients experiencing AEs that resulted in discontinuation of IP during the randomized treatment or follow-up periods was calculated.
Time Frame: Baseline (Week 0) to end of the follow-up period
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NKTR-118 25 mg | Usual Care
Number analyzed (Participants) | 534 | 270
Participants | 56 | NA — Patients in the Usual Care group were not taking any IP and thus could not be categorized for this parameter.

3. Primary Outcome: Incidence of Patients Experiencing Severe Adverse Events (SAEs)
Description: The incidence of patients experiencing SAEs during the randomized treatment and follow-up periods was calculated.
Time Frame: Baseline (Week 0) to end of the follow-up period
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NKTR-118 25 mg | Usual Care
Number analyzed (Participants) | 534 | 270
Participants | 51 | 30

ADVERSE EVENTS:
Arm/Group | NKTR-118 25 mg | Usual Care
Serious Adverse Events (participants affected / at risk) | 51/534 | 30/270
Other Adverse Events (participants affected / at risk) | 365/534 | 152/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 25 mg (N=534) | Usual Care (N=270)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 1 (1)
THYROID MASS (Endocrine disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS OBSTRUCTIVE (Hepatobiliary disorders) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS GANGRENOUS (Infections and infestations) | 1 (1) | 0 (0)
EXTRADURAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 5 (5) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VULVAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD PRESSURE DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 1 (1) | 0 (0)
TROPONIN INCREASED (Investigations) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SUPERFICIAL SPREADING MELANOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
THYROID CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
AKATHISIA (Nervous system disorders) | 1 (1) | 0 (0)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
CERVICAL NEURITIS (Nervous system disorders) | 1 (1) | 0 (0)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
COMPLICATED MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1)
HYPOGLYCAEMIC COMA (Nervous system disorders) | 1 (1) | 0 (0)
IDIOPATHIC GENERALISED EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0)
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
RADICULITIS CERVICAL (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
BIPOLAR I DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
HOMICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
PANIC ATTACK (Psychiatric disorders) | 1 (1) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
SCHIZOPHRENIA (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 2 (2) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 3 (3)
RENAL INJURY (Renal and urinary disorders) | 1 (1) | 0 (0)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 25 mg (N=534) | Usual Care (N=270)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 13 (13) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 12 (12) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 98 (98) | 9 (9)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 30 (30) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 73 (73) | 16 (16)
FLATULENCE (Gastrointestinal disorders) | 39 (39) | 3 (3)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 11 (11) | 5 (5)
NAUSEA (Gastrointestinal disorders) | 56 (56) | 11 (11)
VOMITING (Gastrointestinal disorders) | 28 (28) | 15 (15)
CHILLS (General disorders) | 11 (11) | 0 (0)
FATIGUE (General disorders) | 18 (18) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 13 (13) | 8 (8)
PYREXIA (General disorders) | 14 (14) | 6 (6)
BRONCHITIS (Infections and infestations) | 30 (30) | 12 (12)
GASTROENTERITIS VIRAL (Infections and infestations) | 16 (16) | 4 (4)
INFLUENZA (Infections and infestations) | 10 (10) | 8 (8)
NASOPHARYNGITIS (Infections and infestations) | 33 (33) | 15 (15)
SINUSITIS (Infections and infestations) | 22 (22) | 19 (19)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 31 (31) | 23 (23)
URINARY TRACT INFECTION (Infections and infestations) | 28 (28) | 24 (24)
CONTUSION (Injury, poisoning and procedural complications) | 11 (11) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 19 (19) | 12 (12)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 34 (34) | 16 (16)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 48 (48) | 23 (23)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 17 (17) | 8 (8)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 22 (22) | 7 (7)
DIZZINESS (Nervous system disorders) | 12 (12) | 3 (3)
HEADACHE (Nervous system disorders) | 48 (48) | 13 (13)
ANXIETY (Psychiatric disorders) | 17 (17) | 4 (4)
DEPRESSION (Psychiatric disorders) | 13 (13) | 10 (10)
INSOMNIA (Psychiatric disorders) | 15 (15) | 5 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 8 (8)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 4 (4)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 17 (17) | 1 (1)
HYPERTENSION (Vascular disorders) | 16 (16) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days